CLINICAL TRIAL: NCT01968993
Title: A Prospective, Nonrandomized Study to Assess Lumbar Fusion Using Interbody Cages With Autograft in Conjunction With Instrumented Posterolateral Gutter Fusions Using nanOss Bioactive and Autograft Bone.
Brief Title: Comparison of nanOss Bioactive With Autograft and Bone Marrow Aspirate to Autograft in the Posterolateral Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pioneer Surgical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-02
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis
Keywords: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nanOss Bioactive - posterolateral gutter (Experimental): Participants will undergo instrumented PLF at one or two adjacent levels from L2-S1 with PEEK interbody cages (containing allograft or autograft) using nanOss Bioactive in combination with autograft and bone marrow aspirate in the posterolateral gutter on one side. Autograft alone will be used in the opposite posterolateral gutter.
  Interventions: Device: nanOss Bioactive - posterolateral gutter

INTERVENTIONS:
Device: nanOss Bioactive - posterolateral gutter — Participants will undergo instrumented PLF at one or two adjacent levels from L2-S1 with PEEK interbody cages (containing allograft or autograft) using nanOss Bioactive in combination with autograft and bone marrow aspirate in the posterolateral gutter on one side. Autograft alone will be used in the opposite posterolateral gutter.

SUMMARY:
nanOss Bioactive is approved for use in the U.S. The purpose of this study is to compare fusion results in the posterolateral spine using nanOss Bioactive mixed with autograft bone and bone marrow aspirate (BMA) on one side and autograft alone on the opposite side of the treated level(s). It is hypothesized that the use of nanOss Bioactive will result in fusion at 12 months, with CT evidence of bridging trabecular bone, less than 3mm of translational motion, and less than 5 degrees of angular motion.

DETAILED DESCRIPTION:
The post market clinical investigation is designed to assess instrumented posterolateral fusion (PLF) using nanOss Bioactive bone void filler with autograft bone and bone marrow aspirate in patients with symptomatic spinal stenosis secondary to degenerative disc disease with up to Grade 1 spondylolisthesis at one or two adjacent levels from L2-S1.

Preoperatively, the participant will provide his/her medical history and complete self assessment forms. The investigator will perform a clinical evaluation and x-rays will be performed if recent x-rays are not available. Participants will undergo instrumented PLF with an interbody fusion device (with autograft or allograft) using nanOss Bioactive in combination with autograft bone and bone marrow aspirate in one posterolateral gutter and autograft alone in the opposite posterolateral gutter.

Following surgery, operative and discharge information will be collected and a clinical evaluation will be performed prior to discharge. Participants will be evaluated 6 and 12 months postoperatively. One investigational site will participate in long-term followup of 24 months. Each participant will complete x-rays and self assessment documents. A CT scan performed at the 12 month postoperative visit will be evaluated by an independent radiologist to assess fusion results. Complication data will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* is at least 18 years of age and skeletally mature.
* must have symptomatic spinal stenosis and/or spondylolisthesis or degenerative disc disease (DDD) at one or two adjacent levels from L2-S1 requiring a fusion.
* must have completed a minimum of three months of unsuccessful conservative, non-operative care.
* must have discogenic back pain with or without leg pain.
* DDD must be confirmed by MRI or CT scans followed by discography (if necessary).
* must score at least 40% on the Oswestry Disability Index.
* must score at least a 4 on a 10 cm Visual Analog Scale for back pain.
* must be able to comply with the protocol's follow-up schedule.
* must understand and sign the informed consent document.

Exclusion Criteria:

* symptomatic at more than 2 levels.
* previous fusion surgery at any lumbar level with or without instrumentation (prior discectomy, laminotomy, laminectomy or nucleolysis at the operative (involved) level > 6 months is permitted).
* more than 50% spondylolisthesis.
* lumbar scoliosis greater than 11 degrees.
* osteoporosis, osteopenia, osteomalacia, Paget's disease or metabolic bone disease.
* spinal tumors.
* active arachnoiditis.
* fractures of the epiphyseal plate or fractures for which stabilization of the fracture is not possible.
* impaired calcium metabolism.
* active infection or surgical site infection.
* rheumatoid arthritis or other autoimmune disease
* chronic steroid use (used steroids for one month within the last 6 months) or any medical condition that requires treatment with drugs known to interfere with bone healing.
* systemic disease such as AIDS, HIV, hepatitis (active), tuberculosis.
* morbid obesity defined as body mass index (BMI)>40 or a weight more than 100lbs over ideal body weight.
* smokers unless the patient agrees to quit at least 2 weeks prior to and for the duration of the study, confirmed by a carboxyhemoglobin test prior to surgery.
* psychosocial disorders that would preclude accurate evaluation or has a history of substance abuse.
* active malignancy except non-melanoma skin cancer; history of any invasive malignancy unless treated and in remission for at least five years.
* documented allergies to porcine collagen or titanium
* pregnancy, or interested in becoming pregnant in the next four years.
* participation in another investigational study within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Fusion | 12 months
  Based on x-ray and CT scan. Defined as bridging trabecular bone and less than 3mm of translational motion and less than 5mm of angular motion. X-rays obtained at 6 months and 12 months. CT obtained at 12 months.

SECONDARY OUTCOMES:
Improvement in Oswestry Disability Index score | Preoperatively, 6 months, 12 months
  As compared to baseline levels
Improvement in VAS pain scores | Preoperatively, 6 months, 12 months
  As compared to baseline levels.
Improvement in Short Form-36 scores (SF-36) | Preoperatively, 6 months, 12 months
  As compared to baseline levels.
Decrease in medication usage | Preoperatively, 6 months, 12 months
  As compared to baseline levels.
Work status | Preoperatively, 6 months, 12 months
  As compared to baseline levels.
Patient satisfaction | Preoperatively, 6 months, 12 months
  As compared to baseline levels.

OTHER OUTCOMES:
Complications, adverse events and neurological status | 6 months, 12 months
  Incidence of reoperations, revisions, supplemental fixations, neurological failures, unexpected adverse events or complications will be calculated. Percentage of patients in each category will be reported and exact 95% confidence intervals will be calculated using the inverse beta distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Eastlack, MD, Principal Investigator — Scripps Green Hospital; Thomas Highland, MD, Principal Investigator — Columbia Orthopedic Group
Locations (3):
- United States (3):
  - Scripps Green Hospital, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Columbia Orthopedic Group, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No